CLINICAL TRIAL: NCT05012696
Title: Postextubation Non-invasive Ventilation Versus High-flow Nasal Cannula in Critically Ill Patients At High Risk of Weaning Failure: a Physiologic Randomized Crossover Study
Brief Title: Physiological Effects of Non-invasive Mechanical Ventilation Versus High-flow Nasal Cannula in Critically Ill Patients At High Risk of Extubation Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 210301011
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Weaning from Mechanical Ventilation
Keywords: Noninvasive ventilation; High-flow nasal cannula
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Analysis of work of breathing and of data derived from Electric impedance tomography will be performed blind to arm assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A: Non-invasive ventilation - High flow nasal cannula (Experimental): Once participants are extubated they will receive one hour of Non-invasive ventilation followed by one hour of high-flow nasal cannula.
  Interventions: Device: Non-invasive ventilation (NIV); Device: High-flow nasal cannula
- Sequence B: High flow nasal cannula - Non-invasive ventilation (Experimental): Once participants are extubated they will receive one hour of high flow nasal cannula followed by one hour of Non-invasive ventilation
  Interventions: Device: Non-invasive ventilation (NIV); Device: High-flow nasal cannula

INTERVENTIONS:
Device: Non-invasive ventilation (NIV) — Non-invasive ventilation will be provided through a mechanical ventilator (Carina, Dräger) through a facial interface (Fitlife Respironics, Philips). A PEEP level between 5 and 10 cmH2O, minimal pressure-support level of 5 cm H2O targeting a tidal volume around 6 to 8 ml/kg and at the same FiO2 applied during the spontaneous breathing trial.
Device: High-flow nasal cannula — High flow nasal cannula will be provided through a commercial device (AIRVO2 + Optiflow nasal cannula, Fisher & Paykel), at 50 LPM and at the same FiO2 applied during the spontaneous breathing trial.

SUMMARY:
Weaning is one of the most complex challenges in mechanically ventilated patients. Increased work of breathing after extubation would play a central role in weaning failure. Currently, non-invasive ventilation (NIV) is recommended to prevent weaning failure in high-risk patients. On the other hand, high-flow nasal cannula (HFNC), which is a novel system capable of administering gas mixtures (air and oxygen) with a flow of up to 60 liters/min, has been used to prevent weaning failure in this kind of patients. The use of NIV and HFNC after extubation has been evaluated in some clinical studies. However, the evidence is controversial, and the information regarding the physiological effects that each therapy induces in recently extubated patients at high risk of weaning failure is lacking.

The goal of this proposal is to compare the acute physiological effects of postextubation NIV versus HFNC in critically ill patients at high risk of weaning failure on relevant mechanisms related to weaning failure: Work of breathing, lung function, ventilation distribution, systemic hemodynamics.

This will be a randomized crossover study that will include critically ill mechanically ventilated patients, who fulfill criteria indicating they may be ready for weaning from mechanical ventilation, and in whom a spontaneous breathing trial (SBT) is planned to determine if they should be extubated. After checking eligibility and obtaining informed consent, patients will be monitored with an esophageal catheter (esophageal/gastric pressures to determine work of breathing, and electric activity of diaphragm to determine neuromechanical coupling), and a noninvasive ventilation monitor (electric impedance tomography to assess global and regional ventilation). Work of breathing, lung function, and systemic hemodynamics will be assessed during the SBT. Inclusion in the study will be confirmed only if they pass the SBT and are extubated. During the first 2 hours after extubation, patients will undergo one hour of NIV and one hour of HFNC, with the crossover sequence being randomized previously at the time of inclusion and with assessments repeated at the end of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Mechanical ventilation (MV) through an orotracheal tube for at least 48 hours
2. PaO2 /FiO2 ratio ≤ 300 mmHg (during the MV period)
3. Potential for weaning

   * Precipitating cause leading to MV in resolution
   * PaO2 /FiO2 ratio ≥ 150 mmHg
   * PEEP ≤ 8 cmH2O
   * pH > 7,25
   * SpO2 ≥ 90% with FiO2 ≤ 0.4; BPM ≤35
   * Hemodynamic stability (noradrenaline ≤ 0.1mcg / kg / min and SBP 90-160; HR <140)
   * Temperature <38 ° C
   * Presence of inspiratory effort and appropriate spontaneous cough
   * Decision to perform a spontaneous breathing trial by the attending physician
4. High risk of weaning failure defined by a history of: (i) Previous failed extubation, (ii) Chronic heart or respiratory failure, or (iii) MV ≥ 7 days.

Exclusion Criteria:

1. Contraindications to NIV or HFNC, which include abnormalities, trauma or surgery of the face or nose.
2. Contraindications for esophageal balloon catheter insertion (eg. severe coagulopathy, esophageal varices, and history of esophageal or gastric surgery)
3. Contraindication for use of electric impedance tomography (eg. Pacemaker)
4. Tracheostomy
5. Refusal to participate by the attending physician
6. Do not resuscitate order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Pressure time-product (PTP) per minute | 60 minutes after starting Non-invasive ventilation or high flow nasal cannula
  Pressure time-product (PTP) per minute (cmH2O x s/min)
Esophageal pressure swings (ΔPes) | 60 minutes after starting Non-invasive ventilation or high flow nasal cannula
  Esophageal pressure swings (ΔPes) defined as the absolute differences between end-expiratory and end-inspiratory Pes
End-expiratory lung impedance (EELI) | 60 minutes after starting Non-invasive ventilation or high flow nasal cannula
  End-expiratory lung impedance (EELI)assessed with Electric impedance tomography

SECONDARY OUTCOMES:
Pressure time-product per breath | 60 minutes after starting Non-invasive ventilation or high flow nasal cannula
  Pressure time-product per breath (cmH2O x s). PTP will be assessed through an esophageal Neurovent catheter.
Peak electric activity of the diaphragm (EAdi) | 60 minutes after starting Non-invasive ventilation or high flow nasal cannula
  Peak electric activity of the diaphragm (EAdi) EAdi will be measured in uV through a Neurovent catheter connected to a Servo-i ventilator
Neuroventilatory efficiency | 60 minutes after starting Non-invasive ventilation or high flow nasal cannula
  Neuroventilatory efficiency is a parameter derived from the EAdi signal and the ventilation
Diaphragmatic neuromuscular coupling | 60 minutes after starting Non-invasive ventilation or high flow nasal cannula
  Diaphragmatic neuromuscular coupling Pdi/EAdi
Global inhomogeneity index | 60 minutes after starting Non-invasive ventilation or high flow nasal cannula ]
  Index derived from EIT and calculated from the sum of the impedance changes of each pixel with respect to its median (in absolute values), divided by the sum of the impedance values of each pixel
PaO2 / FiO2 ratio | 60 minutes after starting Non-invasive ventilation or high flow nasal cannula
  Parameter of oxygen exchange calculated as the ratio of PaO2 / FiO2
PaCO2 | 60 minutes after starting Non-invasive ventilation or high flow nasal cannula
  Arterial partial pressure of CO2 (PaCO2) Parameter of alveolar ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico UC Christus, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rochwerg B, Brochard L, Elliott MW, Hess D, Hill NS, Nava S, Navalesi P Members Of The Steering Committee, Antonelli M, Brozek J, Conti G, Ferrer M, Guntupalli K, Jaber S, Keenan S, Mancebo J, Mehta S, Raoof S Members Of The Task Force. Official ERS/ATS clinical practice guidelines: noninvasive ventilation for acute respiratory failure. Eur Respir J. 2017 Aug 31;50(2):1602426. doi: 10.1183/13993003.02426-2016. Print 2017 Aug. PMID 28860265
- [Background] Thille AW, Muller G, Gacouin A, Coudroy R, Decavele M, Sonneville R, Beloncle F, Girault C, Dangers L, Lautrette A, Cabasson S, Rouze A, Vivier E, Le Meur A, Ricard JD, Razazi K, Barberet G, Lebert C, Ehrmann S, Sabatier C, Bourenne J, Pradel G, Bailly P, Terzi N, Dellamonica J, Lacave G, Danin PE, Nanadoumgar H, Gibelin A, Zanre L, Deye N, Demoule A, Maamar A, Nay MA, Robert R, Ragot S, Frat JP; HIGH-WEAN Study Group and the REVA Research Network. Effect of Postextubation High-Flow Nasal Oxygen With Noninvasive Ventilation vs High-Flow Nasal Oxygen Alone on Reintubation Among Patients at High Risk of Extubation Failure: A Randomized Clinical Trial. JAMA. 2019 Oct 15;322(15):1465-1475. doi: 10.1001/jama.2019.14901. PMID 31577036
- [Background] Hernandez G, Vaquero C, Colinas L, Cuena R, Gonzalez P, Canabal A, Sanchez S, Rodriguez ML, Villasclaras A, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation on Reintubation and Postextubation Respiratory Failure in High-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1565-1574. doi: 10.1001/jama.2016.14194. PMID 27706464
- [Background] Mauri T, Turrini C, Eronia N, Grasselli G, Volta CA, Bellani G, Pesenti A. Physiologic Effects of High-Flow Nasal Cannula in Acute Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2017 May 1;195(9):1207-1215. doi: 10.1164/rccm.201605-0916OC. PMID 27997805